CLINICAL TRIAL: NCT03582969
Title: High Intensity, Multi-Donor, Oral Capsulized Fecal Microbiota Transplantation in Newly Diagnosed Pediatric Patients With Mild to Moderate Ulcerative Colitis - a Double Blind, Placebo-Controlled Trial
Brief Title: Capsulized Fecal Microbiota Transplantation in Pediatric Ulcerative Colitis Patients
Acronym: FMT UC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Dr. Ilan Youngster, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0134-17-ASF
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Ulcerative Colitis
Keywords: IBD; UC; fecal-transplantation; capsules; microbiota; microbiome; colitis; pediatric
MeSH Terms: conditions — Colitis, Ulcerative; Colitis | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: This is a placebo-controlled, double blinded interventional study evaluating oral, fecal microbiota transplantation, administered in patients with mild-moderate UC.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The placebo capsules are blocked capsules containing a mixture of saline and glycerine, identical in appearance and consistency to the FMT capsules.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal transplantation (Experimental): Fecal transplantation of feces from healthy donor via capsules. Oral application.
  Interventions: Other: Fecal transplantation
- Placebo (Placebo Comparator): Placebo capsules
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Fecal transplantation — Fecal transplantation administered orally via frozen capsules.
  Arms: Fecal transplantation
Other: Placebo — Placebo capsules
  Arms: Placebo

SUMMARY:
Fecal Microbiota Transplantation(FMT) - reconstitution of normal flora by a stool transplant from a healthy individual, is increasingly being recognized as a therapeutic modality for diseases that are associated with gut dysbiosis.

This is a placebo-controlled, double blinded interventional study evaluating multiple, oral, fecal microbiota transplantation, administered in newly diagnosed pediatric patients with mild-moderate UC.

The primary objective is to assess the safety and feasibility of multiple, oral, fecal microbiota transplantation, in newly diagnosed pediatric patients with mild-moderate UC.

All processing will occur at the Center for Microbiome Research at Assaf Harofeh Medical Center, under GMP conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed (>9 months) with mild to moderate ulcerative colitis as per colonic biopsy and clinical disease activity (SCCAI 5-12).
* Patients not started on immune-suppressive or anti-inflammatory medications (Mesalamine is allowed).
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Women of childbearing potential will have a urine pregnancy test, which must be negative, on Study Day 1, prior to receiving FMT. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study and for 3 months after FMT.
* Ability to understand and the willingness to sign a written document, including the willingness to accept risk of unrelated donor stool.
* Ability of parents or other legal guardian to understand and the willingness to sign a written informed consent document, including the willingness to accept risk of unrelated donor stool.
* Ability to swallow oral medications.

Exclusion Criteria:

* Severe, uncontrolled ulcerative colitis.
* At time of enrollment, immune-suppressive or anti-inflammatory medications, except Mesalamine.
* Patients with active or uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
* Delayed gastric emptying syndrome
* Known chronic aspiration
* Patients with a history of significant allergy to foods not excluded from the donor diet (excluded foods are tree nuts, peanuts, shellfish, eggs)
* Pregnant and breast-feeding women
* Participants who are unable to swallow pills.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
UC remission | 12 weeks
  UC remission at week 12 defined as a Simple Clinical Colitis Activity Index<3

SECONDARY OUTCOMES:
Improvement in UC symptoms | 12 weeks
  defined as improvement in SCCAI
markers of inflammation | 12 weeks, 6 months and 12 months
  Laboratory markers of inflammation - CRP, WBC, ANC, stool calprotectin
Improvement in UC endoscopic score | 12 weeks, 6 months and 12 months
  Mayo-score
change in gut microbiome | 12 weeks, 6 and 12 months.
  Diversity and variability of gut microbiome
use of treatments for UC | 6+12 months
  such as glucocorticoids, immunosuppressive therapy (eg, azathioprine), or tumor necrosis factor antagonists.
Extra-intestinal disease manifestations | 6 and 12 month
  Extra-intestinal disease manifestations

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf-HarofehMC, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Drekonja D, Reich J, Gezahegn S, Greer N, Shaukat A, MacDonald R, Rutks I, Wilt TJ. Fecal Microbiota Transplantation for Clostridium difficile Infection: A Systematic Review. Ann Intern Med. 2015 May 5;162(9):630-8. doi: 10.7326/M14-2693. PMID 25938992
- [Background] Li SS, Zhu A, Benes V, Costea PI, Hercog R, Hildebrand F, Huerta-Cepas J, Nieuwdorp M, Salojarvi J, Voigt AY, Zeller G, Sunagawa S, de Vos WM, Bork P. Durable coexistence of donor and recipient strains after fecal microbiota transplantation. Science. 2016 Apr 29;352(6285):586-9. doi: 10.1126/science.aad8852. PMID 27126044
- [Background] Rossen NG, MacDonald JK, de Vries EM, D'Haens GR, de Vos WM, Zoetendal EG, Ponsioen CY. Fecal microbiota transplantation as novel therapy in gastroenterology: A systematic review. World J Gastroenterol. 2015 May 7;21(17):5359-71. doi: 10.3748/wjg.v21.i17.5359. PMID 25954111
- [Background] Khoruts A, Sadowsky MJ. Understanding the mechanisms of faecal microbiota transplantation. Nat Rev Gastroenterol Hepatol. 2016 Sep;13(9):508-16. doi: 10.1038/nrgastro.2016.98. Epub 2016 Jun 22. PMID 27329806
- [Background] Drekonja D, Reich J, Gezahegn S, Greer N, Shaukat A, MacDonald R, Rutks I, Wilt T. Fecal Microbiota Transplantation for Clostridium Difficile Infection: A Systematic Review of the Evidence [Internet]. Washington (DC): Department of Veterans Affairs (US); 2014 Jul. Available from http://www.ncbi.nlm.nih.gov/books/NBK299000/ PMID 26042318
- [Background] Scaldaferri F, Pecere S, Petito V, Zambrano D, Fiore L, Lopetuso LR, Schiavoni E, Bruno G, Gerardi V, Laterza L, Pizzoferrato M, Ianiro G, Stojanovic J, Poscia A, Papa A, Paroni Sterbini F, Sanguinetti M, Masucci L, Cammarota G, Gasbarrini A. Efficacy and Mechanisms of Action of Fecal Microbiota Transplantation in Ulcerative Colitis: Pitfalls and Promises From a First Meta-Analysis. Transplant Proc. 2016 Mar;48(2):402-7. doi: 10.1016/j.transproceed.2015.12.040. PMID 27109966
- [Background] Moayyedi P, Surette MG, Kim PT, Libertucci J, Wolfe M, Onischi C, Armstrong D, Marshall JK, Kassam Z, Reinisch W, Lee CH. Fecal Microbiota Transplantation Induces Remission in Patients With Active Ulcerative Colitis in a Randomized Controlled Trial. Gastroenterology. 2015 Jul;149(1):102-109.e6. doi: 10.1053/j.gastro.2015.04.001. Epub 2015 Apr 7. PMID 25857665
- [Background] Rossen NG, Fuentes S, van der Spek MJ, Tijssen JG, Hartman JH, Duflou A, Lowenberg M, van den Brink GR, Mathus-Vliegen EM, de Vos WM, Zoetendal EG, D'Haens GR, Ponsioen CY. Findings From a Randomized Controlled Trial of Fecal Transplantation for Patients With Ulcerative Colitis. Gastroenterology. 2015 Jul;149(1):110-118.e4. doi: 10.1053/j.gastro.2015.03.045. Epub 2015 Mar 30. PMID 25836986
- [Background] Youngster I, Russell GH, Pindar C, Ziv-Baran T, Sauk J, Hohmann EL. Oral, capsulized, frozen fecal microbiota transplantation for relapsing Clostridium difficile infection. JAMA. 2014 Nov 5;312(17):1772-8. doi: 10.1001/jama.2014.13875. PMID 25322359
- [Background] Kelly CR, Ihunnah C, Fischer M, Khoruts A, Surawicz C, Afzali A, Aroniadis O, Barto A, Borody T, Giovanelli A, Gordon S, Gluck M, Hohmann EL, Kao D, Kao JY, McQuillen DP, Mellow M, Rank KM, Rao K, Ray A, Schwartz MA, Singh N, Stollman N, Suskind DL, Vindigni SM, Youngster I, Brandt L. Fecal microbiota transplant for treatment of Clostridium difficile infection in immunocompromised patients. Am J Gastroenterol. 2014 Jul;109(7):1065-71. doi: 10.1038/ajg.2014.133. Epub 2014 Jun 3. PMID 24890442
- Available data/document: Clinical Study Report — https://www.ncbi.nlm.nih.gov/pubmed/25938992